CLINICAL TRIAL: NCT03131518
Title: From Cars to Bikes - the Feasibility and Effect of Using E-bikes, Traditional Bikes and Longtail Bikes for Transportation Among Parents of Children Attending Kindergarten: a Randomized Cross-over Trial
Brief Title: From Cars to Bikes - the Feasibility and Effect of Bicycling for Transportation Among Parents of Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Agder (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); The National Association for Public Health, Norway (Other Government)
Responsible Party: Principal Investigator, Helga Birgit Bjørnarå, Postdoctoral Research Fellow, University of Agder
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1320 98842
Record Dates: First submitted 2017-04-19; First posted 2017-04-27 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Bicycling Distance; Bicycling Time; Physical Activity Level; Cardiorespratory Fitness; Body Composition

STUDY DESIGN:
Intervention Model Description: All participants in the intervention group (n=18) will complete the following intervention arms in random order: (i) 3 months access to an e-bicycle with trailer (n=6), (ii) 3 months access to a longtail bicycle (n=6), and (iii) 3 months access to a regular bicycle with trailer (n=6), in total 9 months. Also, a control group (n=18) maintaining usual transportation and PA habits will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-bicycle (Other): Access to an e-bicycle will be provided.
  Interventions: Behavioral: Access to an e-bicycle with trailer
- Longtail bicycle (Other): Access to a longtail bicycle will be provided.
  Interventions: Behavioral: Access to a longtail bicycle
- Traditional bicycle (Other): Access to a traditional bicycle will be provided.
  Interventions: Behavioral: Access to a traditional bike with trailer

INTERVENTIONS:
Behavioral: Access to an e-bicycle with trailer — Participants will be provided with an e-bike with trailer for 3 months.
  Arms: E-bicycle
Behavioral: Access to a longtail bicycle — Participants will be provided with a longtail bike for 3 months.
  Arms: Longtail bicycle
Behavioral: Access to a traditional bike with trailer — Participants will be provided with a traditional bicycle with trailer for 3 months.
  Arms: Traditional bicycle

SUMMARY:
There is a need for a greater understanding of e-bikes and their role in the transportation network, and further effects on physical activity (PA) levels and health. Moreover, longtail bikes could meet certain practical needs not sufficiently fulfilled by e-bikes or traditional bikes, hence increased knowledge regarding their potential and feasibility should be obtained. No intervention study has investigated whether providing an e-bike or a longtail bike over an extended period in a sample of inactive parents of toddlers influence objectively assessed amount of cycling, total PA level, potential mode shifts, and effect on cardiorespiratory fitness, body composition and blood pressure.

Objectives:

To assess the effect of an intervention where participants have access to an e-bike (including a trailer), a longtail bike and a traditional bike (including a trailer) on the following parameters:

1. Objectively assessed amount of biking, total levels of PA, and mode shifts from car/motorized modes to bicycle.
2. Cardiorespiratory fitness, blood pressure, body composition, self-reported health and health-related quality of life (HRQoL).
3. Experiences with bicycling (el/longtail/traditional) and intrinsic motivation for bicycling.
4. How season and weather conditions influence the amount of bicycling (el/longtail/traditional).

Study sample:

A convenience sample consisting of 36 inactive parents of toddlers will be recruited among residents in Kristiansand municipality, Southern Norway.

Measures:

The following measures will be conducted:

1. A web-based questionnaire will assess socio-demographics (at baseline only), transportation habits, self-perceived health and HRQoL, and motivation for bicycling for transportation. For the intervention group: at baseline and post all intervention arms, i.e. four times. For the control group: at baseline and after 9 months, i.e. two times.
2. Cycling time and distance will be assessed through usage of a cycle computer throughout the entire project period, in total nine months.
3. Time spent in moderate-to-vigorous PA (MVPA) will be estimated with the monitor SenseWear Armband Mini (SWA) for seven consecutive days at study start and after 9 months (post-intervention).
4. Cardiorespiratory fitness will be measured performing treadmill walking/running, and dual-energy X-ray absorptiometry (DXA) will be used for assessing body composition. In addition, blood pressure, body weight and height (height only at baseline) will be measured at baseline and after 9 months (post-intervention).
5. Participants' experiences with and motivation for usage of the different bicycle types will be explored in semi-structured focus group interviews after 3 months, 6 months and 9 months.
6. Weather data (temperature, rainfall, snow, etc.) will also be collected.

Scientific contribution:

The present study will add knowledge to relevant and topical areas, i.e. issues related to public health and environmental sustainability, among parents of toddlers, representing an important target group.There is a call for research on the influence of e-bikes on travel behavior and level of MVPA, and whether voluntary cycling with e-bikes could improve health. Moreover, to our knowledge no scientific studies have assessed possible effects of using a longtail bike, on the selected parameters. If the current study reveals promising results, it should be replicated in a larger and more representative sample of parents of toddlers, as well as in other important target groups (e.g. older adults). If findings are positive, inclusion in national public health policies should be considered.

ELIGIBILITY:
Inclusion Criteria:

* being able to understand and read Norwegian
* having one child born in 2013, 2014 or 2015 attending kindergarten
* being responsible for bringing/picking up the "study child" in the kindergarten ≥5 times per week/at least half of the times
* residing 2-10 km from the workplace
* residing <3 km from the kindergarten and the grocery shop
* having car-access
* possessing a smartphone
* being between 167-190 cm tall (due to the size of accessible bicycles)
* having the opportunity to store the bicycles indoors

Exclusion Criteria:

* having bicycled more than once weekly during the last 12 months to either the workplace, the kindergarten, or the grocery shop.
* suffering from severe cardiovascular diseases or upper respiratory tract diseases.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Amount of bicycling | In total 9 months, 3 months for each bicycle type.
  Bicycling distance and time will be combined to assess change in total amount of bicycling for transportation.

SECONDARY OUTCOMES:
Physical activity level | 2 weeks; one week at baseline, and one week after 9 months (post-intervention).
  Change in total time of MVPA.
Cardiorespiratory fitness | Baseline and 9 months (post-intervention).
  Change in VO2 max.
Body composition | Baseline and 9 months (post-intervention).
  Change in body composition.
Blood pressure | Baseline and 9 months (post-intervention).
  Change in blood pressure.

OTHER OUTCOMES:
Feasibility and motivation for bicycling (qualitative) | Retrospective after 3 months, 6 months and 9 months (post-intervention).
  Experiences with bicycling for transportation, and changes in motivation for bicycling for transportation.

CONTACTS AND LOCATIONS:
Overall Officials: Elling Bere, Prof., Principal Investigator — University of Agder
Locations (1):
- University of Agder, Kristiansand, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjornara HB, Berntsen S, Te Velde SJ, Fegran L, Fyhri A, Deforche B, Andersen LB, Bere E. From cars to bikes - the feasibility and effect of using e-bikes, longtail bikes and traditional bikes for transportation among parents of children attending kindergarten: design of a randomized cross-over trial. BMC Public Health. 2017 Dec 28;17(1):981. doi: 10.1186/s12889-017-4995-z. PMID 29282108